CLINICAL TRIAL: NCT07165886
Title: Phase II/III Study to Evaluate the Safety and Efficacy of Sirolimus for Injection (Albumin Bound) Combined With Octreotide Long-acting Injection in Patients With Metastatic Gastroenteropancreatic Neuroendocrine Tumors (GEP-NETs)
Brief Title: Sirolimus for Injection (Albumin Bound) Combined With Octreotide Long-acting Injection in Patients With Metastatic Gastroenteropancreatic Neuroendocrine Tumors
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HB1901-010
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumors
MeSH Terms: interventions — Sirolimus; Injections; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sirolimus combined with octreotide (Experimental): Sirolimus for injection (albumin bound) combined with octreotide long-acting injection (Q2W) will be administrated on a 28-day cycle
  Interventions: Drug: Sirolimus for injection (albumin bound); Drug: Octreotide long-acting injection
- Sirolimus monotherapy (Experimental): Sirolimus for injection (albumin bound) (Q2W) will be administrated on a 28-day cycle.
  Interventions: Drug: Sirolimus for injection (albumin bound)
- Everolimus monotherapy (Active Comparator): Everolimus (QD) will be orally administrated on a 28-day cycle. Only for Phase III
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Sirolimus for injection (albumin bound) — Sirolimus for injection (albumin bound), ivgtt., Q2W
  Arms: Sirolimus combined with octreotide; Sirolimus monotherapy
Drug: Octreotide long-acting injection — SC, Q2W
  Arms: Sirolimus combined with octreotide
Drug: Everolimus — Oral, once a day
  Arms: Everolimus monotherapy

SUMMARY:
There is limited evidence regarding the benefit of adding somatostatin analogs to molecular targeted agents for well-differentiated gastroenteropancreatic neuroendocrine tumors (GEP-NETs) with poor prognostic factors. This trial was conducted to evaluate sirolimus for injection (albumin bound) combined with octreotide long-acting injection in patients with unresectable or recurrent GEP-NETs in the first-line setting.

ELIGIBILITY:
Inclusion Criteria:

* 1. Unresectable locally advanced or metastatic G1/G2 GEP-NETs diagnosed by histology, according to the 2019 WHO histological grading criteria.
* 2. Have not received systemic anti-tumor treatment for neuroendocrine tumors in the past.
* 3. Having poor prognostic factors.
* 4. Non-functional GEP-NETs are required.
* 5. At least one measurable lesion that meets the RECIST V1.1 standard.
* 6. ECOG 0~2.
* 7. Organ function reserve is good.
* 8. Be able to sign a written informed consent form.

Exclusion Criteria:

* 1. Received treatment with other unlisted clinical investigational drugs within 4 weeks prior to the first use of the investigational drug.
* 2. Undergone major surgical procedures within 4 weeks prior to the first use of the investigational drug and have not fully recovered.
* 3. Received systemic use of corticosteroids or other immunosuppressive therapy within 2 weeks prior to the first use of the study drug.
* 4. With an infection that requires systemic anti-infective treatment within 2 weeks prior to the first use of the study drug.
* 5. Those who have used strong inhibitors or inducers of CYP3A4 liver metabolic enzymes within 2 weeks prior to the first use of the investigational drug or still need to continue using such drugs.
* 6. Has a serious history of cardiovascular and cerebrovascular diseases.
* 7. Having active brain metastasis and/or malignant meningitis.
* 8. With a history of severe lung diseases.
* 9. During screening, there may be symptomatic gallstones or a history of symptomatic gallstones but no surgical treatment has been performed.
* 10. Abnormal thyroid function during screening.
* 11. Known to have hypersensitivity reactions or intolerance to any component of all investigational drugs or their excipients.
* 12. Active hepatitis B, active hepatitis C virus infection, or active syphilis infection.
* 13. History of autoimmune diseases (excluding tuberous sclerosis), history of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2028-08-29 (Estimated); Study Completion 2028-08-29 (Estimated)

PRIMARY OUTCOMES:
Phase II: Incidences of Adeverse Events (AEs) | Up to 3 years
Phase II: Maximum tolerated dose (DLT) | Up to 1 year
Phase II: Recommended Phase 3 Dose (RP3D) | Up to 1 year
Phase II: Objective Response Rate (ORR） per investigator | Up to 1 year
Phase III: Progression Free Survival (PFS) per Independent Review Committee (IRC) | Up to 3 years

SECONDARY OUTCOMES:
Phase II: Duration of Response (DOR) per investigator | Up to 3 years
Phase II: Disease Control Rate (DCR) per investigator | Up to 3 years
Phase II: Progression Free Survival (PFS) per investigator | Up to 3 years
Phase II/III: Overall Survival (OS) | Up to 3 years
Peak Concentration：Cmax | Up to 3 years
Area under the plasma concentration-time curve: AUC | Up to 3 years
Half-Life: t1/2 | Up to 3 years
Phase III: Progression Free Survival (PFS) per investigator | Up to 3 years
Phase III: Objective Response Rate (ORR） | Up to 3 years
Phase III: Duration of Response (DOR) | Up to 3 years
Phase III: Disease Control Rate (DCR) | Up to 3 years
Phase III: Incidences of Adeverse Events (AEs) | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China